CLINICAL TRIAL: NCT00894842
Title: A 10-week, Randomized, Double-Blind, Placebo-Controlled Trial of a Neurocognition Enhancing Agent(Pregnenolone) in Patients With Schizophrenia.
Brief Title: Study of a Neurocognition Enhancing Agent in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Research Foundation, Singapore (Other Government)
Collaborators: Duke University (Other); National University of Singapore (Other); Singapore Clinical Research Institute (Other)
Responsible Party: Principal Investigator, Chong Siow Ann, Associate Professor, National Research Foundation, Singapore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCR-NS-003
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Pregnenolone; Neurocognition
MeSH Terms: conditions — Schizophrenia | interventions — Pregnenolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregnenolone (Active Comparator)
  Interventions: Drug: Pregnenolone
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregnenolone — Pregnenolone 50 mg BID x 14 days, followed by Pregnenolone 300 mg per day for 14 days (200 mg qAM and 100 mg qPM), followed by Pregnenolone 500 mg per day for the remainder of the 8-week trial (300 mg qAM and 200 mg qPM)
  Arms: Pregnenolone
Drug: Placebo — Placebo 50 mg BID x 14 days, followed by Placebo 300 mg per day for 14 days (200 mg qAM and 100 mg qPM), followed by Placebo 500 mg per day for the remainder of the 8-week trial (300 mg qAM and 200 mg qPM)
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to determine whether pregnenolone will demonstrate significant improvements in cognitive functioning and negative symptoms compared to patients receiving placebo.

DETAILED DESCRIPTION:
Aims:

Schizophrenia is one of the most disabling disorders to afflict mankind. Despite the low lifetime prevalence of schizophrenia (1% world-wide), it has an enormous burden in both economic cost and human suffering. There is currently no cure for schizophrenia and its cause is not well understood. Patients with schizophrenia also suffer from negative symptoms (loss of drive, apathy, poverty of speech) and severe cognitive impairments especially with memory, attention, processing of information - the latter of which is most robustly correlated with their role functioning in the community. Addressing these impairments with effective interventions is thus critically important but at this present moment, there is no effective treatment. Recent emerging data from animal studies and a pilot study on small group of patients with schizophrenia suggest that neurosteroids such as pregnenolone may be relevant to schizophrenia pathophysiology and treatment of neurocognitive impairments. This study will be a 10-week randomised double-blind placebo-controlled trial of the efficacy and safety of pregnenolone. Our hypothesis is patients with schizophrenia randomized to pregnenolone will demonstrate significant improvements in cognitive functioning and negative symptoms compared to patients receiving placebo. The primary aims of the study are to demonstrate the efficacy of pregnenolone in comparison to placebo in patients with schizophrenia which are assessed by changes (from baseline) in the composite score of the MATRICS Consensus Cognitive Battery (MCCB), BACS and the Scale for Assessment of Negative Symptoms (SANS). Changes in functionality will be assessed by the University of California Performance Based Skills Assessment (UPSA). Safety will be assessed with laboratory tests, well established scales for side effects as well as with a side-effects checklist.

Objectives:

To demonstrate the efficacy of pregnenolone in comparison to placebo in patients with schizophrenia and with cognitive impairment from randomization (Week 2) to Week 10 by using MATRICS Consensus Cognitive Battery, BACS, Scale for Assessment of Negative Symptoms, Performance Based Skills Assessment - Brief Version and Clinical Global Impression -Improvement (CGI-I).Additional safety data on pregnenolone in patients with schizophrenia will be provided.

Methodology:

The proposed study is a single-site, randomized, double blind placebo-controlled comparison of adjunctive pregnenolone and placebo. A total sample will consist of 120 clinically stable inpatients and outpatients with DSM IV schizophrenia, with 60 subjects randomized to each group. A best estimate diagnostic approach will be utilized, in which information from the Structured Clinical Interview for DSM-IV will be supplemented by information from family informants, previous psychiatrists, and medical records to generate a diagnosis. There will be a 2 week, single-blind placebo lead-in evaluation phase, in which subjects will undergo baseline diagnostic and medical testing, including a physical examination, Electrocardiogram (ECG), Complete Blood Counts (CBC), complete metabolic panel, urine toxicology, and urinalysis. The study is designed to confirm the pilot study results (n=9 per group; total of 18 patients of 21 randomized who completed at least 4 weeks of treatment) in a larger clinical trial (n=60 per group, 120 patients total). Identical to our pilot study, patients will be seen for a total of 6 study visits (every two weeks). The placebo arm is essential as there are no standard therapies for cognitive defects as yet.

Potential Benefits:

While patients may not personally be helped by taking part in this study, their participation may lead to knowledge that will help better understand the illness. It may also lead to better treatment for cognitive deficits and negative symptoms in schizophrenia.

Potential Risks:

Obtaining blood can cause pain, bleeding, bruising, or swelling at the site of the needle prick. There is a risk that some questions on the questionnaires might upset the patients or cause psychological distress. There are no known severe risks that had been associated with taking pregnenolone.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 21 to 65 years inclusively at screening.
* Current diagnosis of Schizophrenia established by Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for at least 1 year prior to screening.
* Subjects can be either inpatients or outpatients.
* Provision of written informed consent.
* Able to understand and comply with the requirements of the study, as judged by the investigator.
* Subjects have to be treated with a first generation and/or second generation antipsychotic for the previous 8 weeks or longer, with no change in dose in ≥ 4 weeks at screening.
* Women of childbearing potential (less than two years post-menopausal or not surgically sterile), must have a negative urine pregnancy test at screening - and must use a highly effective method of birth control for at least one month prior to screening such as barrier methods, implants, sexual abstinence or vasectomised partner.

Exclusion Criteria:

* Subjects with a DSM-IV diagnosis of alcohol or other substance dependence (other than nicotine) within the last month.
* Subjects with a history of significant head injury/trauma, with loss of consciousness (LOC) for more than 1 hour, recurring seizures resulting from the head injury, clear cognitive sequelae of the injury, or cognitive rehabilitation following the injury.
* Subjects with a history of clinically significant neurological, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, and/or urological disorders (e.g., unstable angina, seizures, cerebrovascular accident, decompensate congestive heart failure, CNS infection, HIV seropositivity), which would pose a risk to the patient if they were to participate in the study or that might confound the results of the study.

  * Active medical conditions that are minor or well-controlled are not exclusionary if they are not likely to affect risk to the patient or the study results.
  * Patients with hormone-sensitive tumours (such as breast, uterine, or prostate cancer) will be excluded.
* Clinically significant abnormalities in physical examination, ECG, or laboratory assessments.
* Pregnant women or sexually active women of child-bearing potential, who are either not surgically-sterile or not using appropriate methods of birth control (urine pregnancy test will be performed at baseline and week 10 of the study to exclude pregnancy).
* Women who are breast-feeding.
* ECT treatment within the last 3 months.
* Use of oral contraceptives or other hormonal supplementation such as oestrogen.
* Subjects who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others.
* Known allergy to study medication.
* Participation in another drug trial within 4 weeks of this study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Improvement in composite score of the MATRICS Consensus Cognitive Battery (MCCB) and BACS. | 10 weeks
Improvement of negative symptoms as assessed by the Scale for Assessment of Negative Symptoms (SANS). | 10 weeks

SECONDARY OUTCOMES:
To provide additional safety data on pregnenolone in patients with schizophrenia via reported serious and non serious adverse events. | 10 weeks
Improvement of functional outcome by the University of California Performance Based Skills Assessment (UPSA-B)at Week 2, 6 and 10. | 10 weeks
Efficacy outcome variables will be evaluated by the Clinical Global Impression -Improvement (CGI-I) score at week 2 to week 10. | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Siow Ann Chong, Principal Investigator — Vice Chairman of Medical Board (Research)
Locations (1):
- Institute of Mental Health, Singapore, Singapore